CLINICAL TRIAL: NCT03846908
Title: Postprandial Lipid Metabolism in Patients With Hypertriglyceridemia and Normo-lipidemic Controls: Medium Chain Fatty Acids (MCT) in Comparison to Long-chain, Saturated Fatty Acids (SFA) and Mono-unsaturated Fatty Acids (MUFA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Klaus Parhofer, Professor of Endocrinology and Metabolism, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: MCT-HTG
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MCT (Experimental): subjects start with MCT fat load
  Interventions: Other: MCT; Other: SFA; Other: MUFA
- SFA (Experimental): subjects start with SFA fat load
  Interventions: Other: MCT; Other: SFA; Other: MUFA
- MUFA (Experimental): subjects start with MUFA fat load
  Interventions: Other: MCT; Other: SFA; Other: MUFA

INTERVENTIONS:
Other: MCT — patients will receive fat load with MCT
Other: SFA — patients will receive fat load with SFA
Other: MUFA — patients will receive fat load with MUFA

SUMMARY:
Postprandial lipid metabolism will be evaluated in patients with hypertriglyceridemia and normo-lipidemic controls; different fats will be used (saturated fatty acids, mon-unsaturated fatty acids and medium chain fatty acids) for the oral fat challenge.

ELIGIBILITY:
Inclusion Criteria:

* hypertriglyceridemia (150 mg/dl-900 mg/dl)

Exclusion Criteria:

* Lipid lowering drugs or indication for Lipid lowering drugs
* LDL-cholesterol > 190 mg/dl
* Diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
postprandial hypertriglyceridemia | 8 hours after fat meal
  area under the curve following oral fat load

CONTACTS AND LOCATIONS:
Locations (1):
- University Munich, Munich, Germany